CLINICAL TRIAL: NCT05590949
Title: Post-menopausal Breast Cancer Patients Treated With Aromatase Inhibitors and Denosumab: An Observational Study to Assess Rebound Bone Loss and Insufficiency Fractures After Denosumab Discontinuation
Brief Title: Observational Study of Bone Complications in People With Post-menopausal Breast Cancer Who Have Stopped Treatment With Denosumab and Aromatase Inhibitors
Status: Recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 22-280
Record Dates: First submitted 2022-10-18; First posted 2022-10-21 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer
Keywords: Post-menopausal Breast Cancer; Breast Cancer; Denosumab; Aromatase; 22-280; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Breast Neoplasms | interventions — Absorptiometry, Photon

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Post- menopausal breast cancer patients: Participants are post- menopausal with a breast cancer diagnosis who received at least 2 doses of denosumab, and then discontinued therapy, and discontinued Aromatase Inhibitors/AI prior to or within 6 months of stopping denosumab
  Interventions: Other: Physical Evaluation; Diagnostic Test: Dual-energy X-ray absorptiometry scans; Diagnostic Test: Trabecular Bone Score

INTERVENTIONS:
Other: Physical Evaluation — Participants will be assessed at Timepoint 0 (last dose of denosumab injection) and then at 9,12,18 and 24 months following discontinuation of denosumab. The evaluation will include history and pain assessment for development of new fractures, weight and height measurement with BMI (body mass index) calculation, and blood work for bone turnover markers (including serum carboxy-terminal collagen crosslinks (CTX) in serum and bone specific alkaline phosphatase). Bone turn-over markers should be drawn in the morning, after at least 8 hours of fasting (water, black coffee and plain tea allowed).
Diagnostic Test: Dual-energy X-ray absorptiometry scans — Dual-energy X-ray absorptiometry (DEXA) scans will be performed at the 12 months timepoint , and then at the 24 month timepoint.
  Other Names: DEXA scans
Diagnostic Test: Trabecular Bone Score — TBS is an innovative gray-level texture measurement that utilizes lumbar spine DEXA images to discriminate changes in bone microarchitecture. Specifically, TBS measures bone quality through tridimensional bone areas with different trabecular and microstructural characteristics. The combination of TBS microstructure evaluation with bone density measured by DEXA has been shown to be superior to either measurement alone in the assessment of fracture risk.
  Other Names: TBS

SUMMARY:
The purpose of this study to gather information about changes in the bones after stopping treatment with aromatase inhibitor/AI and denosumab. The study team will collect information from 5 standard clinic visits over the course of 24 months. The information will include information about participant health assessments, blood test results, and imaging results. After 24 months, participation in this study will be complete.

ELIGIBILITY:
Inclusion Criteria:

* Women with confirmed diagnosis of breast cancer
* Participant must be post-menopausal, defined as last menstrual cycle at least 12 months prior to enrollment
* Received at least 2 doses of denosumab and then discontinued therapy
* Discontinued AI prior to or within 6 months of last denosumab injection
* Patients must be 18 years of age or olde

Exclusion Criteria:

* Patients with history of osteoporosis prior to starting denosumab, based on previous dual-energy X-ray absorptiometry (DEXA) scan;
* Patients with history of insufficiency fracture.
* Patients who continue treatment with a different bone modifying agent (i.e oral or intravenous bisphosphonates) after discontinuation of denosumab
* Patients on chronic low-dose glucosteroids.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited through the Breast Medicine and Survivorship Services. Members of the research team will verify eligibility against the patient's medical record. Once eligibility is confirmed, and if the treating investigator has no objection to enrolling the patient in the research study, the patient will be approached for consent. Consent to the protocol will be conducted by a trained consenting professional. Consent will take place either in the clinic, or by following the most updated standard working procedures for consent via telemedicine.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-10-18 (Actual); Primary Completion 2026-10-18 (Estimated); Study Completion 2026-10-18 (Estimated)

PRIMARY OUTCOMES:
Change in serum carboxy-terminal collagen crosslinks (CTX) | 12 months
  Evaluate changes in bone turnover markers at 12 months after the last dose of denosumab - serum carboxy-terminal collagen crosslinks (CTX)
Change in bone specific alkaline phosphatase (ALK) | 12 months
  Evaluate changes in bone turnover markers at 12 months after the last dose of denosumab - bone specific alkaline phosphatase (ALK)

CONTACTS AND LOCATIONS:
Overall Officials: Monica Fornier, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk-Commack (Limited protocol activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org